CLINICAL TRIAL: NCT03077490
Title: Comparison of Single Versus Multicenter Outcomes for Pelvic Organ Prolapse Repair Using a Mesh-capturing Device
Acronym: KIDS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Edward Morcos, Senior consultant, MD, PhD, Karolinska Institutet
Other Study IDs: Protokoll Dnr 2015/5: 3
Record Dates: First submitted 2017-02-01; First posted 2017-03-13 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Prolapse Genital
Keywords: Pelvic organ prolapse; transvaginal mesh; complications
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single center vs. multicenter: Both Groups operated on by the same device (Transvaginal mesh Uphold TM Vaginal Support System) and in the same manner.
  Interventions: Device: Transvaginal mesh Uphold TM Vaginal Support System; Device: Transvaginal mesh Uphold TM Vaginal Support System.

INTERVENTIONS:
Device: Transvaginal mesh Uphold TM Vaginal Support System
  Other Names: Transvaginal mesh Uphold TM Vaginal Support System.
Device: Transvaginal mesh Uphold TM Vaginal Support System.

SUMMARY:
Comparison of single versus multicenter outcomes for pelvic organ prolapse repair using a mesh-capturing device (The Uphold™ Vaginal Support System for apical and vaginal wall prolapse - Boston Scientific). 1-2 years follow up study comprison of 112 vs 207 patients.

DETAILED DESCRIPTION:
112 women operated by two surgeons at one center (2 years follow up) are to be compared to 207 women operated by twenty six surgeons at twenty four centers (1 year follow-up).

Screening at baseline for apical (uterine or vaginal vault) prolapse stage II with or without concomitant anterior or vaginal wall prolapse ≥ stage 2 according to the pelvic organ prolapse quantification (POP-Q) system.

Surgical data including operation data, complications and hospital stay are to be compared.

Anatomical outcome measurements by POP-Q evaluations. Subjective symptoms are to be evaluated by prolapse specific symptom questionnaires (PFIQ-7, UDI-6 and PFIQ) whereas sexual function to be estimated by PISQ-12.

ELIGIBILITY:
Inclusion

* Posthysterectomy prolapse of the vaginal apex, with or without cystocele, where the vaginal apex descends at least 50% of the total vaginal length
* Uterine prolapse, with or without cystocele, where the leading edge of the cervix descends at least 50% of the total vaginal length and TVL minus point C= ≤ 2 cm
* Prolapse specific pelvic symptom of pelvic heaviness and/or vaginal bulging
* Reproductive years in the past (biologically or reproductive decision)
* Being able to make an informed consent on participation
* Physically and cognitively capable of participating in the required follow-up
* No exclusion criteria fulfilled

Exclusion Criteria:

* Posthysterectomy prolapse of the vaginal apex where the vaginal apex descends less than 50% of the total vaginal length regardless of whether a cystocele is present or not
* Uterine prolapse, with or without cystocele, where the leading edge of the cervix descends less than 50% of the total vaginal length
* If cervix elongation is present corresponding to: TVL minus point C= >2 cm.
* If prolapse specific pelvic symptoms of pelvic heaviness and/or vaginal bulging are not present
* Previous or current pelvic organ cancer (regardless of treatment)
* Severe rheumatic disease
* Insulin treated diabetes mellitus
* Connective tissue disorders (SLE, Sjögrens syndrome, Marfans syndrome, Ehlers Dahnlos, collagenosis, polymyositis eller rheumatic myalgia)
* Current systemic steroid treatment
* Other clinically relevant pelvic disorders for which surgery is indicated including stress urinary incontinence, cervix elongation and posterior prolapse
* Decision to perform prolapse surgery using other medical devices/mesh

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 112 patients from single center compared to 207 patients from 24 different centers
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
The rate of immediate complications | From operation start to hospital discharge, assessed for an estimated total of days (1-7 days).
  Serious surgical complications are categorized as any surgical event which is potentially life-threatening related to the surgical procedure including: internal organ perforation (or other injury), bleeding in excess of 1000 mL.
Rate of delayed complications | From hospital discharge and up to 2 years at single center and 1 year at multicenter
  Adverse events during follow-up which requires re-hospitalisation or surgical re-intervention.

SECONDARY OUTCOMES:
Anatomical outcomes | 2 years vs 1 year
  Anatomical outcome is a composite definition including point C positioned above a point corresponding to half of the total vaginal length. The overall POP-Q outcomes will be analyzed to determine efficacy of the procedure related to correction of anterior prolapse ≥stage II or other defects present at the time of surgery. Days in hospital are counted from the day of surgery i.e. the day of operation is day 1 and the day of returning home is the last day of hospital stay.
Subjective outcomes and sexual function | 2 years vs 1 year
  Subjective outcome is the patients' response 'no' to question 2 of the PFDI (pelvic heaviness). The composite outcome is a strictly binary categorization where any residual sense of pelvic heaviness/vaginal bulging results in the classification of the patient as a failure. It also includes the components of the main secondary outcome considered individually, any adverse events in the aftermath of surgery, as well as, patient-reported urogenital distress (UDI), quality of life (PFIQ) and sexual function (PISQ-12) as measured by the self-reported questionnaires. For secondary analyses, the ordinal grading of responses to the PFDI-20, PFIQ-7 and PISQ-12 will be used to determine rates of improvement and progression over time.
Ultrasound mapping of mesh position in the pelvic floor and correlation to anatomical and subjective outcomes and sexual function | 5, 7, 10 years
  Mesh measurements: Total mesh midsagittal length, length above and below the bladder neck (BN) level. Distance between mesh lower edge and pubis symphysis (PS) lower edge and PS level.
  Bladder neck: Distance between BN and PS levels. Distance between BN and PS lower edge.
  Urethra: Total urethra length. Distance between mid-urethra and PS lower edge and PS level.
  Using identical examination protocol, independent examination at rest and physical strain is to be done by senior gynecologist at an ultrasound referral unit and gynecologist. Estimation of intra class coefficient (ICC) in-between examiners in order to determine method reproducibility.
  To statistically compare between the collected ultrasound data and clinical outcomes. Clinical outcomes include anatomical, subjective and sexual function outcome.
Measurement of Pain by patient self-reporting Visual analogue scale (VAS-scale) | Changes from baseline, 2, 5 and 10 years after surgery
  VAS scale is a numeric rating scale and ranges from 0-10 (each digit is 1cm) where 0 indicates no and 10 indicates maximum, digits between 0-10 indicate degree of pain.
Measurement of urinary incontinence by patient self-reporting Visual analogue scale (VAS-scale) | Changes from baseline, 2, 5 and 10 years after surgery
  VAS scale is a numeric rating scale and ranges from 0-10 (each digit is 1cm) where 0 indicates no and 10 indicates maximum, digits between 0-10 indicate degree of severity of urinary incontinence. VAS scale for urinary incontinence: 0 indicate no urinary incontinence whereas 10 indicates maximal or severe urinary incontinence.
Measurement of patient satisfaction by patient self-reporting Visual analogue scale (VAS-scale) | assessment at 2, 5 and 10 years after surgery
  VAS scale is a numeric rating scale and ranges from 0-10 (each digit is 1cm) where 0 indicates no and 10 indicates maximum, digits between 0-10 indicate degree of satisfaction after mesh surgery. VAS scale for patient satisfaction: 0 indicates no satisfaction whereas 10 indicates maximal satisfaction.
12. Measurement of patient recommendation to other patients to undergo same surgery with vaginal mesh if they suffer apical prolapse, assessed by patient self-reporting Visual analogue scale (VAS-scale) | assessment at 2, 5 and 10 years after surgery
  VAS scale is a numeric rating scale and ranges from 0-10 (each digit is 1cm) where 0 indicates no and 10 indicates maximum, digits between 0-10 indicate degree of satisfaction. VAS scale for patient recommendation to other patients to undergo same surgery if they suffer apical prolapse: 0 indicates no recommendation whereas 10 indicates maximal recommendation.

IPD SHARING:
Plan to Share IPD: No